CLINICAL TRIAL: NCT02659371
Title: Weight Loss by Low Energy Diet as Treatment Prior Mamma Reduction in Overweight Women - A Pilot Study
Brief Title: Weight Loss Prior Mamma Reduction - A Pilot Study
Acronym: MAMMARED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen University Hospital at Herlev (Other)
Responsible Party: Principal Investigator, Christian Bitz, Head of research, Copenhagen University Hospital at Herlev
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EFFECT.C02.2014
Record Dates: First submitted 2015-11-09; First posted 2016-01-20 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Weight Loss; Hypertrophy
MeSH Terms: conditions — Weight Loss; Hypertrophy | interventions — Caloric Restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Low energy diet (Experimental): Low energy diet (800 kcal/d) for eight weeks, following 4 weeks on reintroduction supplying 1200 kcal/d.
  Interventions: Dietary Supplement: Low energy diet

INTERVENTIONS:
Dietary Supplement: Low energy diet

SUMMARY:
Due to a higher risk of complications, obese and overweight patients with macromastia are in Denmark prohibited mammoplasty , as BMI must be within normal range, i.e. BMI < 25 kg/m2.

The study is a pilot study with a diet intervention group and no control group. The intervention is a 12 week low energy diet pre-operative weight loss program investigating if this will result in weight loss making the overweight and obese patients eligible for breast reduction surgery i.e. BMI < 25.

ELIGIBILITY:
Inclusion Criteria:

* entitled to mammoplasty,
* motivated towards participation in a weight loss program
* BMI within the range 25.5 to 35 kg/m2

Exclusion Criteria:

* more than 65 years of age
* insulin-dependent diabetes
* chronic heart, liver or kidney failure

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-01; Primary Completion 2015-01 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Weight loss | 12 weeks
  Measurement of weight to nearest 0.1 kg on category III approved body weight

SECONDARY OUTCOMES:
Breast volumen | 12 weeks
  measure of breast volumen
Breast size | 12 weeks
  anthropometric measurements of the breasts by measuring tape.
Pain and discomfort | 12 weeks
  Questionnaire on pain in head, neck, shoulders

OTHER OUTCOMES:
Blood bio markers | 12 weeks
  Blood sampling and analyses of blood bio markers, e.g. lipids
Hip circumference | 12 weeks
  Measurements of hip circumference to nearest 0.1 cm by measuring tape, repeated three times.
Waist circumference | 12 weeks
  Measurements of waist circumference to nearest 0.1 cm by measuring tape, repeated three times.

CONTACTS AND LOCATIONS:
Overall Officials: Arne Astrup, MDDrMedSci, Principal Investigator — University of Copenhagen
Locations (1):
- Copenhagen University Hospital at Herlev (EFFECT), Herlev, Herlev, Denmark